CLINICAL TRIAL: NCT02468154
Title: Efficacy of Leg Casts With Heel Off-loaded in Children: Open Randomized Controlled Trial
Brief Title: Efficacy of Leg Casts With Heel Off-loaded in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 79/14
Record Dates: First submitted 2014-11-24; First posted 2015-06-10 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2015-09

CONDITIONS: Orthopedic Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- splint (Experimental): Splint is placed under the cast of children affected by spasticity who have to keep the heel unloaded.
  Interventions: Device: custom made splint
- standard care (Active Comparator): To avoid pressure at the heel placing and maintaining the limb with the cast on cushions or folded sheets so that the heel is not resting on the bed plane
  Interventions: Other: standard off-load plaster cast

INTERVENTIONS:
Device: custom made splint — Splints have been made by wrapping synthetic bandages around a leg-foot manufactured splint padded at the heel to off-load the heel. When the desired shape has been obtained, the splint is opened and the manufactured device is removed, thus obtaining a device that is used under the casts of lower limbs.
  Arms: splint
Other: standard off-load plaster cast — To avoid pressure at the heel placing and maintaining the limb with the cast on cushions or folded sheets so that the heel is not resting on the bed plane
  Arms: standard care

SUMMARY:
Assess whether by placing a "custom made" splint with heel in the immediate postoperative period until removal of the cast, the rate of pain, the number of healthcare interventions to maintain the off-loaded heel position and number of pressure sores in children wearing lower limb plaster casts is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Treated by operations to the lower limbs which require immediate plaster casts that include the foot
* Treated by osteotomy, joint fusion, patella repositioning and fracture fixation
* Children with intact skin at the heel

Exclusion Criteria:

* Caregivers who cannot speak Italian
* Those who refuse to give their consent to take part in the study
* Patients with lower limb casts that are allowed to load the limb

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Veronesi, RN, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2014-August 2015, 57 paediatric orthopaedic patients who need a lower limb plaster cast after surgery out of the 172 potentially eligible (33.1%) were enrolled in the trial.
Period: Overall Study
Arm/Group | Splint | Standard Care
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Splint | Standard Care | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.96) | 10.5 (3.72) | 10.5 (3.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  Italy | 29 | 28 | 57
bone surgical intervention (vs soft tissue surgical intervention) [Number; unit: participants] | 22 | 21 | 43
spica cast [Number; unit: participants] | 9 | 4 | 13
over the knee cast [Number; unit: participants] | 11 | 16 | 27
under the knee cast [Number; unit: participants] | 9 | 8 | 17
pain killer (opioid) [Number; unit: participants] | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain Score on the "Numeric Rating Scale" or "Visual Rating Scale" or "Face, Legs Activity Cry Consolability" According to Age Group
Description: All scales had values from 0 to 10 where zero represented no pain and 10 the worst possible pain
Time Frame: up to the first 2 days during hospitalization and at cast removal (maximum 30 days).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Splint | Standard Care
Number analyzed (Participants) | 29 | 28
units on a scale | 4.4 (2.4) | 3.9 (3)

2. Secondary Outcome: Numbers of Participants With Heel Pressure Sores Detected According to the Classification of the Scale of the National Pressure Ulcer Advisory Panel -N.P.U.A.P.
Time Frame: one time at cast removal (expected average of 30 days).
Measure: Number; unit: participants
Arm/Group | Splint | Standard Care
Number analyzed (Participants) | 29 | 28
participants | 1 | 5

3. Secondary Outcome: Health Staff/Caregiver Interventions
Description: daily number of interventions by health staff /caregiver to maintain the cast in an off-loaded position, marked on a form given daily to the family/caregiver
Time Frame: up to the first 2 days during hospitalization
Measure: Mean (Standard Deviation); unit: daily number of interventions
Arm/Group | Splint | Standard Care
Number analyzed (Participants) | 29 | 28
daily number of interventions | 2.1 (3.2) | 5.2 (3.6)

4. Secondary Outcome: Comfort Perceived by the Patient and by the Caregiver Using a Scale of 0 to 10
Description: The scales had values from 0 to 10 where zero represented no comfort perceived and 10 the best comfort perceived
Time Frame: one time at cast removal (expected average of 30 days).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Splint | Standard Care
Number analyzed (Participants) | 29 | 28
units on a scale | 8.9 (1.1) | 7.6 (1.7)

ADVERSE EVENTS:
Arm/Group | Splint | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes